CLINICAL TRIAL: NCT05437250
Title: A French Multicentric Observational Study of Acalabrutinib in the Treatment of Chronic Lymphocytic Leukemia Patients
Brief Title: National Acalabrutinib Observational Study
Acronym: NAOS
Status: Active, not recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D8220R00045
Record Dates: First submitted 2022-06-08; First posted 2022-06-29 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- CLL patients treated with acalabrutinib at their physician's discretion: In each center, all patients meeting the inclusion criteria and no exclusion criteria will be offered to participate in this study.
  Interventions: Drug: Non interventional study

INTERVENTIONS:
Drug: Non interventional study — CLL patients initiated with acalabrutinib at their physician's discretion between January 1, 2021 and December 31, 2022 . Secondary data collection

SUMMARY:
The efficacy and safety of acalabrutinib in the treatment of patients with chronic lymphocytic leukemia (CLL) have been well established through 3 phase III clinical trials (ELEVATE TN, ASCEND, ELEVATE R/R) that led to European Medicines Agency approval in November 2020. The aim of this French longitudinal, non-interventional/observational, multicenter study is to describe the efficacy and safety of acalabrutinib treatment for CLL patients in real life.

The primary objective is then to estimate the time to discontinuation of acalabrutinib therapy and the reasons for discontinuation, overall and by treatment line.

The secondary objectives are to describe the baseline clinical and demographic characteristics of patients with CLL treated with acalabrutinib, to assess the efficacy of acalabrutinib through progression-free survival, overall survival, time to next treatment or death, describe acalabrutinib treatment patterns in CLL patients and reasons, identify key determinants of acalabrutinib discontinuation in CLL patients, estimate healthcare resource utilization. The overall response rate will be estimated as an exploratory objective.

Patients included in this study will be CLL patients treated with acalabrutinib at the discretion of their physician between January 1, 2021 and December 31, 2022, who have been informed of the study and do not object to electronic processing of their data for research purposes (or do not object during their lifetime in the event of the patient's death prior to study initiation).

Secondary data will be extracted from the hospital's patient records once a year. The protocol calls for the recruitment of 350 patients at 70 centres with a 3-year follow-up. Interim analyses will be performed annually until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥ 18 years old,
* CLL patients initiated with acalabrutinib at their physician's discretion between January 1st 2021 and December 31st 2022,
* Patients alive at study initiation and who have been informed verbally and/or in writing about this study, and who do not object to their data being electronically processed or subjected to data quality control (certified by physician); or patient who died before study initiation and who did not object to data collection for research purpose(s) during his or her lifetime.

Exclusion Criteria:

* Patients participating in a clinical trial with an investigational drug within 30 days prior to acalabrutinib initiation,
* Patients who initiated acalabrutinib treatment before January 1st 2021.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CLL patients
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2022-09-13 (Actual); Primary Completion 2026-11-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Time to Discontinuation | Up to 3 years from the start of acalabrutinib
  Time between first day of acalabrutinib and the day that acalabrutinib is stopped

SECONDARY OUTCOMES:
Baseline clinical and demographic characteristics in CLL patients | First interim analysis (year1) and second interim analysis (year2)
  Demographic characteristics (gender, age BMI) and disease characteristics (age at diagnosis, previous treatment, staging, prognosis criteria, constitutive symptoms)
Effectiveness of acalabrutinib | Once a year until end of study (up to 3 years from the start of acalabrutinib)
  Real World Progression Free Survival Overall Survival Time to next treatment or Death
Major determinants of treatment discontinuation | Once a year until end of study (up to 3 years from the start of acalabrutinib)
  Multivariate analysis to study correlation between Time to Discontinuation and patient characteristics at baseline
Acalabrutinib interruption | Once a year until end of study (up to 3 years from the start of acalabrutinib)
  Percentage of patients with acalabrutinib interruption
Reasons of acalabrutinib interruption | Once a year until end of study (up to 3 years from the start of acalabrutinib)
  Reasons of acalabrutinib interruption
Time to interruption | Once a year until end of study (up to 3 years from the start of acalabrutinib)
  Time between first day of acalabrutinib and the day of first interruption of acalabrutinib
Duration interruption | Once a year until end of study (up to 3 years from the start of acalabrutinib)
  Time between first day of acalabrutinib interruption and the day of acalabrutinib restart
Acalabrutinib dose changes | Once a year until end of study (up to 3 years from the start of acalabrutinib)
  Percentage of patients with acalabrutinib dose changes
Reasons of Acalabrutinib dose changes | Once a year until end of study (up to 3 years from the start of acalabrutinib)
  Reasons of acalabrutinib dose changes
Healthcare Resources Utilization : Hospitalization | Once a year until end of study (up to 3 years from the start of acalabrutinib)
  Number of day of hospitalization
Healthcare Resources Utilization : Accident and Emergency Visits | Once a year until end of study (up to 3 years from the start of acalabrutinib)
  Number of Accident and Emergency Visits
Healthcare Resources Utilization : Outpatient Visits | Once a year until end of study (up to 3 years from the start of acalabrutinib)
  Number of Outpatient Visits

OTHER OUTCOMES:
Overall Response Rate | Once a year until end of study (up to 3 years from the start of acalabrutinib)
  Response to treatment assessed by investigator

CONTACTS AND LOCATIONS:
Overall Officials: Anne Quinquennel, Doctor, Study Director — Hôpital Robert Debré, Reims, France
Locations (61):
- France (61):
  - Research Site, Aix-en-Provence
  - Research Site, Amiens
  - Research Site, Angers
  - Research Site, Ars-Laquenexy
  - Research Site, Avignon
  - Research Site, Besançon
  - Research Site, Béziers
  - Research Site, Bobigny
  - Research Site, Bourg-en-Bresse
  - Research Site, Brest
  - Research Site, Caen
  - Research Site, Cahors
  - Research Site, Carcassonne
  - Research Site, Cesson-Sévigné
  - Research Site, Chalon-sur-Saône
  - Research Site, Chambéry
  - Research Site, Clamart
  - Research Site, Clermont-Ferrand
  - Research Site, Corbeil-Essonnes
  - Research Site, Dunkirk
  - Research Site, Essey-lès-Nancy
  - Research Site, Grenoble
  - Research Site, La Chaussée-Saint-Victor
  - Research Site, La Tronche
  - Research Site, LE Chesnay-rocquencourt
  - Research Site, Le Kremlin-Bicêtre
  - Research Site, Le Mans
  - Research Site, Le Puy-en-Velay
  - Research Site, Lens
  - Research Site, Libourne
  - Research Site, Lille
  - Research Site, Limoges
  - Research Site, Lorient
  - Research Site, Marseille
  - Research Site, Meaux
  - Research Site, Melun
  - Research Site, Mont-de-Marsan
  - Research Site, Nantes
  - Research Site, Nevers
  - Research Site, Nîmes
  - Research Site, Orléans
  - Research Site, Paris
  - Research Site, Perpignan
  - Research Site, Pessac
  - Research Site, Périgueux
  - Research Site, Pontoise
  - Research Site, Reims
  - Research Site, Rennes
  - Research Site, Roubaix
  - Research Site, Rouen
  - Research Site, Saumur
  - Research Site, Tarbes
  - Research Site, Toulouse
  - Research Site, Tours
  - Research Site, Trévenans
  - Research Site, Troyes
  - Research Site, Valence
  - Research Site, Vandœuvre-lès-Nancy
  - Research Site, Vantoux
  - Research Site, Vesoul
  - Research Site, Vichy

IPD SHARING:
Plan to Share IPD: No